CLINICAL TRIAL: NCT00219713
Title: A Randomized Placebo-Controlled Double Blind Trial Comparing Pre-Mixed 50 Per Cent Nitrous Oxide and Oxygen Mixture in Combination With Local Local 1% Xylocaine Anesthetic Versus Placebo in Order to Evaluate Pain Intensity During Bone Marrow Biopsy.
Brief Title: Evaluation of Pain Intensity During Bone Marrow Biopsy Performed With Inhalation of Pre-Mixed 50 Per Cent Nitrous Oxide and Oxygen Mixture.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); Air Liquide Santé International (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 991300
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Pain
Keywords: Nitrous oxide and oxygen; Pain; Bone marrow biopsy; Bone marrow aspiration
MeSH Terms: conditions — Pain | interventions — Nitrous Oxide; Oxygen

INTERVENTIONS:
Drug: nitrous oxide and oxygen

SUMMARY:
Bone marrow biopsy is a painful medical procedure often performed with local anesthetic.

Therefore a double-blind, randomized, controlled trial was carried out in 330 adult patients who where referred for bone marrow biopsy and aspiration. 164 were assigned to inhale an equimolar mixture of nitrous oxide and oxygen and 166 to inhale a placebo. Pain measurement used visual-analogue pain scales, which involve rating the intensity of pain on a horizontal ruler

DETAILED DESCRIPTION:
The efficacy of an inhaled equimolar mixture of nitrous oxide and oxygen to prevent procedural pain during lumbar puncture in children has been demonstrated. In adults the use of an inhaled equimolar mixture could prevent pain.

Although nitrous oxide was initially considered innocuous, evidence began to be gathered later that it had potentially side effect. It has been demonstrated that nitrous oxide inactivates the vitamin B12-dependent enzyme methionine synthetase and impairs DNA synthesis in bone marrow cells.

Therefore this prospective, multicenter randomized placebo controlled, double-blind trial was design to determine whether an inhaled equimolar mixture of nitrous oxide and oxygen would significantly reduce pain during bone marrow biopsy with aspiration. In addition we performed a careful cytological examination of bone marrow samples in order to evaluate the quality of the picture sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* with a good clinical condition (score ECOG < 2)
* without contra indication for the use of nitrous oxide or previous medical history of allergy to Xylocaïne.
* Informed consent signed up.

Exclusion Criteria:

* pregnancy,
* prior exposure to nitrous oxide,
* patients with neurological illness and those on anti depressant medications or with congestive heart failure or significant respiratory disease.
* patients on analgesia for other medical conditions or whose with the inability to provided consent of an assessment of pain.
* patients with platelet dysfunction or related coagulation disorders, aspirin or warfarin therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280
Dates: Start 2000-03; Study Completion 2004-12

PRIMARY OUTCOMES:
Reduce pain during bone marrow biopsy with aspiration.

SECONDARY OUTCOMES:
Tolerability
Evaluation of the quality of the picture sample

CONTACTS AND LOCATIONS:
Overall Officials: François GUILHOT, MD, Study Chair — Department of Oncology hematology and Cell therapy, University Hospital , 86021 Poitiers - FRANCE
Locations (1):
- University Hospital, Poitiers, France